CLINICAL TRIAL: NCT06344000
Title: A Study of the Association Between Progression and Nutritional Status in Bronchiectasis
Brief Title: Study on Disease Progression and Nutritional Status in Bronchiectasis
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wang xiaorong, Internal medicine physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: RICU20240323
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Bronchiectasis
Keywords: Nutrition; Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: inapplicable — inapplicable

SUMMARY:
Bronchiectasis is a common lung disease. The Bronchiectasis Severity Index (BSI) is a widely used assessment system. The body mass index (BMI) is a commonly used measure of nutritional status, but it has its limitations. To provide a more comprehensive assessment, the investigators also consider other nutrition-related indices such as upper arm circumference, calf circumference, skinfold thickness and grip strength. The investigators will specify the relationship between nutritional status and disease progression by measuring nutrition-related indicators and tracking participants' disease progression.

DETAILED DESCRIPTION:
Non-cystic fibrosis bronchiectasis is a common lung disease in which low body weight and BMI are in more common. The prevalence of malnutrition is higher in bronchiectasis compared to other lung diseases. A study on the assessment of nutritional status in end-stage lung disease noted a higher prevalence of malnutrition in patients with CF or NCFB according to the GLIM framework. Therefore nutritional status is a condition of concern in patients with non-cystic fibrosis bronchiectasis. The Bronchiectasis Severity Score (BSI), of which BMI is a component, is a useful prognostic measure, and it is reasonable to assume that BMI correlates with the severity of bronchiectasis.BMI is an easily accessible nutrition-related criterion, and many studies have been conducted on the correlation between BMI and prognosis, including hospitalisation, in patients with bronchiectasis. It has been shown that BMI is an independent predictor of hospitalisation and that patients with lower BMI are more likely to have acute exacerbations, worsening lung function, increased systemic inflammation and chronic colonisation by Pseudomonas aeruginosa. It has now been shown that reduced muscle mass in patients with lower nutritional status (especially fat-free mass index) is thought to contribute to worsening lung function in patients with COPD. This phenomenon may still be present in patients with bronchiectasis.BMI, a commonly used body measure in clinical practice, is easy to obtain but does not adequately reflect the nutritional status of the participants, so the researchers included new nutritional parameters such as upper arm circumference, calf circumference, grip strength, skinfold thickness, upper arm muscle circumference, and defatted body mass index in order to comprehensively assess the nutritional status of the patients, and to clarify the relationship between nutritional status and bronchiectasis. correlation between nutritional status and the presence of prognosis in bronchiectasis. According to the inclusion and exclusion criteria, participants with confirmed diagnosis of bronchiectasis attending the Union Hospital of Tongji Medical College of Huazhong University of Science and Technology from 31 March 2024 to 31 March 2027 will be included in this study. At the time of enrolment, the researchers collected the demographic information of the participants such as gender, age, measurement of their height (m), weight (kg), skinfold thickness (including triceps brachii, back, and abdomen) (mm), upper arm circumference (cm), calf circumference (cm), grip strength (average of two measurements in kilograms using a grip strength meter), and data from bioelectrical impedance analysis (phase angle (phA), total fat mass (FM), fat-free mass (FFM), skeletal muscle mass (SMM) ), and blood test results such as red blood cell count (10^12/l), haemoglobin (g/l), triglycerides (mmol/l), LDL cholesterol (mmol/l), HDL cholesterol (mmol/l), and blood glucose (mmol/l) were collected from the participants' blood tests at the time of their visit. The results of pulmonary function tests, such as the patient's FEV1 and FEV1 as a percentage of the expected value, and imaging tests of the lungs, such as CT, were also used to calculate the patient's nutrition-related indices, such as BMI (kg/m^2), fat-free mass index (FFMi), and the patient's nutrition-related indices, such as BMI (kg/m^2) and FFMi (FFMi). free mass index (FFMi) and skeletal muscle mass index (SMMi)), and the participants' PNI index, CONUT index, HALP index, GNRI index, GPS index, and Bhalla Scoring. After enrolment, the participants were grouped into malnourished and non-malnourished groups according to the GLIM criteria based on the nutritional status of the patients. Over the next three years, the patients were followed up every six months to obtain the above nutritional indices, pulmonary function and lung CT results, as well as the number of acute exacerbations, the number of hospitalisations, and the survival status of the patients per year, in order to conclude the relationship between nutritional status and the progression of bronchiectasis.

Methods： Height, weight, upper arm circumference, calf circumference and waist circumference were determined while the patients were fasting and wearing only light clothing. Waist circumference was determined to the nearest 0.1 cm. Waist circumference was measured just above the ilium using flexible plastic measuring tape. Upper arm circumference is measured at the triceps belly. Calf circumference is measured at the quadriceps belly.Body height (in meters) was measured using a normal height scale and body weight was determined using digital devices . BMI was determined using the following formula: body weight in kilograms divided by body height in meters squared.

Handgrip strength was measured on three separate occasions . This was performed with the patient seated on a chair, with their shoulder and forearm in a neutral position and the elbow at 90 degrees of flexion. The participant performed a maximum grip force for 3 s and rested for 1 min between each repetition.

Total fat mass and total fat-free mass were determined via bioelectrical impedance (BIA) analysis with a total accuracy of 50 g. The bioelectrical impedance analysis was performed in a standardized manner, with the patient fasting for 8 h and resting for 30 min. The electrodes were placed distally on the wrists and ankles of the patients, with the patients in a supine position and having assumed a lying position 30 min beforehand. Absolute fat-free mass (FFM) and skeletal muscle mass (SMM) were determined directly via impedance. Then, FFMi (fat-free mass index) was determined by dividing absolute FFM by squared height (FFM (kg)/height (m2)); SMMi (skeletal muscle mass index) was also determined by dividing SMM by squared height. Subjects were separated into 2 groups according to their median SMMi values.

The CONUT score was calculated from the results of three laboratory tests, including serum albumin level, total lymphocyte count and cholesterol level. The calculation formula of the PNI score was as follows: 10∗serum albumin level (g/dL) + 0.005∗ total lymphocyte count (number/mm3). The GNRI score was calculated as 14.89 ∗ serum albumin level (g/dL) + 41.7 ∗ (current weight/ideal weight), and the ideal weight was calculated as 22 ∗ height squared. The HALP score is calculated as HALP Score = [hemoglobin (g/L) * albumin (g/L) *lymphocytes (/L)]/platelets (/L).The Glasgow prognostic score (GPS) is evaluated using serum CRP and albumin levels.Lung CT scores were scored according to the Bhalla scoring criteria and were co-scored by two medical imaging physicians.

Statistical analysis and statistical methods： The data obtained during the study were pre-collated. For continuous data, normality tests were first performed. If all groups met normality, the Student's t-test was used for comparison between groups. Otherwise, the non-parametric Wilcoxon rank sum test was considered. For categorical variables, the χ2 test was used. Statistically significant data were subjected to multivariate logistic regression analysis. Receiver operating characteristic (ROC) and Delong's method were used to analyze the effect of different nutritional status on the prognosis of participants with bronchiectasis，with a difference considered statistically significant at P < 0.05.

Statistical analysis of all data was performed through SPSS (IBM SPSS Statistics 26.0, SPSS Inc., Chicago, IL) and R language (version 4.1.3, www.R-project.org/). All statistical tests were two-sided, and statistical significance was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Participants' pulmonary imaging findings and clinical presentation met the diagnostic criteria for bronchiectasis
* Informed consent was signed

Exclusion Criteria:

* Age <18 years
* Does not meet the diagnostic criteria for bronchiectasis
* Participants with cystic fibrosis or previous lung transplantation
* Participants who are unable to cooperate with the study due to dysfunction of vital systems such as heart, brain, liver, and kidneys, or who are unable to participate in the study due to comorbid serious diseases
* Pregnant or lactating females
* Who are not able to provide informed consent or who refuse to participate in the clinical study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with lung Computed Tomography findings and clinical symptoms consistent with bronchiectasis.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of acute exacerbations of bronchiectasis | From the start of inclusion to one year later.
  Acute exacerbations of bronchiectasis were defined according to the consensus published in the European Journal of Respiratory Sciences in 2017, and the frequency of acute exacerbations per year was obtained from participants through follow-up visits

SECONDARY OUTCOMES:
Deterioration of lung function | From the start of inclusion to one year later.
  Participants obtained FEV1 as a percentage of predicted value from pulmonary function tests and scored pulmonary function according to the Bronchiectasis Severity Scale on a scale of 0-2, with higher scores representing poorer lung function
Severity of dyspnoea | From the start of inclusion to one year later.
  Dyspnoea was graded according to Modification of the UK Medical Research Council Dyspnoea Scale (mMRC), ranging from 0-IV, with higher grades being associated with more severe dyspnoea
Bhalla scores on CT of participants' lungs | From the start of inclusion to one year later
  A Bhalla severity score was performed and recorded on lung CT at enrolment and during annual follow-up. The Bhalla score is 0-25, with higher scores indicating greater severity.
Frequency of hospitalisation | From the start of inclusion to one year later.
  Frequency of hospitalisation for bronchiectasis among participants in a year
Death | From the start of inclusion to one year later.
  Participants died during follow-up because of bronchiectasis as the main cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Wang, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (2):
- China (2):
  - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan Union Hospital,China, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
In this study, we will share parts of the study design such as Study Protocol, Statistical Analysis Plan (SAP) and Informed Consent Form (ICF).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share the data 6 months after the end of the study, which lasts for 3 years
Access Criteria: Data were obtained through the Principal Investigator of this study upon reasonable request.

REFERENCES:
- [Background] Cederholm T, Jensen GL, Correia MITD, Gonzalez MC, Fukushima R, Higashiguchi T, Baptista G, Barazzoni R, Blaauw R, Coats AJS, Crivelli AN, Evans DC, Gramlich L, Fuchs-Tarlovsky V, Keller H, Llido L, Malone A, Mogensen KM, Morley JE, Muscaritoli M, Nyulasi I, Pirlich M, Pisprasert V, de van der Schueren MAE, Siltharm S, Singer P, Tappenden K, Velasco N, Waitzberg D, Yamwong P, Yu J, Van Gossum A, Compher C; GLIM Core Leadership Committee, GLIM Working Group. GLIM criteria for the diagnosis of malnutrition - A consensus report from the global clinical nutrition community. J Cachexia Sarcopenia Muscle. 2019 Feb;10(1):207-217. doi: 10.1002/jcsm.12383. PMID 30920778
- [Background] Calanas-Continente A, Gutierrez-Botella J, Garcia-Curras J, Cobos MJ, Vaquero JM, Herrera A, Molina MJ, Galvez MA. Global Leadership Initiative on Malnutrition-Diagnosed Malnutrition in Lung Transplant Candidates. Nutrients. 2024 Jan 27;16(3):376. doi: 10.3390/nu16030376. PMID 38337661
- [Background] Chalmers JD, Goeminne P, Aliberti S, McDonnell MJ, Lonni S, Davidson J, Poppelwell L, Salih W, Pesci A, Dupont LJ, Fardon TC, De Soyza A, Hill AT. The bronchiectasis severity index. An international derivation and validation study. Am J Respir Crit Care Med. 2014 Mar 1;189(5):576-85. doi: 10.1164/rccm.201309-1575OC. PMID 24328736
- [Background] Despotes KA, Choate R, Addrizzo-Harris D, Aksamit TR, Barker A, Basavaraj A, Daley CL, Eden E, DiMango A, Fennelly K, Philley J, Johnson MM, McShane PJ, Metersky ML, O'Donnell AE, Olivier KN, Salathe MA, Schmid A, Thomashow B, Tino G, Winthrop KL, Knowles MR, Daniels MLA, Noone PG. Nutrition and Markers of Disease Severity in Patients With Bronchiectasis. Chronic Obstr Pulm Dis. 2020 Oct;7(4):390-403. doi: 10.15326/jcopdf.7.4.2020.0178. PMID 33108111
- [Background] Onen ZP, Gulbay BE, Sen E, Yildiz OA, Saryal S, Acican T, Karabiyikoglu G. Analysis of the factors related to mortality in patients with bronchiectasis. Respir Med. 2007 Jul;101(7):1390-7. doi: 10.1016/j.rmed.2007.02.002. Epub 2007 Mar 19. PMID 17374480
- [Background] Qi Q, Li T, Li JC, Li Y. Association of body mass index with disease severity and prognosis in patients with non-cystic fibrosis bronchiectasis. Braz J Med Biol Res. 2015 Aug;48(8):715-24. doi: 10.1590/1414-431X20154135. Epub 2015 Jul 10. PMID 26176309
- [Background] Cao C, Wang R, Wang J, Bunjhoo H, Xu Y, Xiong W. Body mass index and mortality in chronic obstructive pulmonary disease: a meta-analysis. PLoS One. 2012;7(8):e43892. doi: 10.1371/journal.pone.0043892. Epub 2012 Aug 24. PMID 22937118
- [Background] Kwan HY, Maddocks M, Nolan CM, Jones SE, Patel S, Barker RE, Kon SSC, Polkey MI, Cullinan P, Man WD. The prognostic significance of weight loss in chronic obstructive pulmonary disease-related cachexia: a prospective cohort study. J Cachexia Sarcopenia Muscle. 2019 Dec;10(6):1330-1338. doi: 10.1002/jcsm.12463. Epub 2019 Jun 17. PMID 31207189
- [Background] Vestbo J, Prescott E, Almdal T, Dahl M, Nordestgaard BG, Andersen T, Sorensen TI, Lange P. Body mass, fat-free body mass, and prognosis in patients with chronic obstructive pulmonary disease from a random population sample: findings from the Copenhagen City Heart Study. Am J Respir Crit Care Med. 2006 Jan 1;173(1):79-83. doi: 10.1164/rccm.200506-969OC. PMID 16368793
- [Background] Hachisu Y, Murata K, Takei K, Tsuchiya T, Tsurumaki H, Koga Y, Horie T, Takise A, Hisada T. Prognostic nutritional index as a predictor of mortality in nontuberculous mycobacterial lung disease. J Thorac Dis. 2020 Jun;12(6):3101-3109. doi: 10.21037/jtd-20-803. PMID 32642232
- [Background] Miano N, Di Marco M, Alaimo S, Coppolino G, L'Episcopo G, Leggio S, Scicali R, Piro S, Purrello F, Di Pino A. Controlling Nutritional Status (CONUT) Score as a Potential Prognostic Indicator of In-Hospital Mortality, Sepsis and Length of Stay in an Internal Medicine Department. Nutrients. 2023 Mar 23;15(7):1554. doi: 10.3390/nu15071554. PMID 37049392
- [Background] Hill AT, Haworth CS, Aliberti S, Barker A, Blasi F, Boersma W, Chalmers JD, De Soyza A, Dimakou K, Elborn JS, Feldman C, Flume P, Goeminne PC, Loebinger MR, Menendez R, Morgan L, Murris M, Polverino E, Quittner A, Ringshausen FC, Tino G, Torres A, Vendrell M, Welte T, Wilson R, Wong C, O'Donnell A, Aksamit T; EMBARC/BRR definitions working group. Pulmonary exacerbation in adults with bronchiectasis: a consensus definition for clinical research. Eur Respir J. 2017 Jun 8;49(6):1700051. doi: 10.1183/13993003.00051-2017. Print 2017 Jun. PMID 28596426